CLINICAL TRIAL: NCT06770387
Title: Telenursing and Transitional Care After Lumbar Disc Herniation Surgery: A New Paradigm for Postoperative Care
Brief Title: Telenursing and Transitional Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Kadiriye Pehlivan, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: New Paradigma
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Surgery
Keywords: mHealth; telenursing; transitional care; lumbar disc surgery; complications
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): No intervention, only routin care
- Intervention Group (Experimental): Telenursing and mHealth intervention
  Interventions: Behavioral: mhealth

INTERVENTIONS:
Behavioral: mhealth — mobile application for postoperative period
  Arms: Intervention Group

SUMMARY:
Post-operative care for Lumbar Disc Herniation (LDH) is important to reduce postoperative complications. The transition from hospital to home after discharge is important for LDH patients, as the transition process is flawless, the necessary care is provided appropriately, and follow-up is important. The aim of the study is to determine the effects of transitional model-based telenursing and mobile application-based follow-up on fall risk, post-discharge recovery, mobility, anxiety, and complications in patients who underwent lumbar disc surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older,
* Can speak and understand Turkish,
* Have no hearing, understanding, vision or speech problems,
* Have undergone LDH surgery for the first time,
* Have undergone LDH surgery with the open method,
* Have not been diagnosed with depression or anxiety disorder before surgery and are not taking medication for this purpose,
* Have a smart mobile phone suitable for taking photos or for those close to them,
* Have not developed serious complications that would delay their discharge from the hospital,
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Patients who wish to withdraw from the study at any stage after voluntarily participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Complication | From enrollment to the end of treatment at 1 weeks
  developing complications
Rehospitalization | From enrollment to the end of treatment at 1 weeks
  hospitalization in the postoperative period
Readmission | From enrollment to the end of treatment at 1 weeks
  admission to hospital in the postoperative period

SECONDARY OUTCOMES:
Measuring recovery status with the Post-Discharge Surgical Recovery Scale | From enrollment to the end of treatment at 4 weeks
  Postoperative recovery
mobilization | From enrollment to the end of treatment at 4 weeks
  postoperative mobilization
Measurement of anxiety status with the hospital anxiety depression scale | From enrollment to the end of treatment at 4 weeks
  Determination of change in anxiety levels between groups before discharge and one month after discharge

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Deva Hospital, Gaziantep
  - Gaziantep University Şahinbey Research and Application Hospital, Gaziantep
  - Medical Point Hospital, Gaziantep
  - Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No